CLINICAL TRIAL: NCT07147309
Title: Multimodal PET Imaging With 18F-FDG/SV2A/TSPO for Resection Planning in Drug-Resistant Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Weibing Miao, PhD (Other)
Responsible Party: Sponsor-Investigator, Weibing Miao, PhD, professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: FirstAHFujian-2504
Record Dates: First submitted 2025-08-19; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; PET / MR; Synaptic Vesicle Proteins; Microglial Activation; FDG PET
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focuses on the application value of 18F-FDG, SV2A, and TSPO PET imaging in the preoperative localization of epileptogenic foci in epilepsy. 18F-FDG PET detects glucose metabolism in brain tissue and is characterized by reduced metabolism during the interictal period. It is currently the most commonly used localization method in clinical practice, especially suitable for temporal lobe epilepsy, but has limited sensitivity to foci with insignificant metabolic changes. SV2A PET targets synaptic vesicle proteins and reflects synaptic density, showing reduced uptake in epileptogenic foci areas. It has high localization accuracy, can effectively supplement the diagnosis of 18F-FDG PET-negative cases, and also has good application prospects in non-temporal lobe epilepsy. TSPO PET monitors microglial activation to reflect neuroinflammation, with increased uptake in epileptogenic foci areas, and has unique auxiliary diagnostic value in refractory epilepsy and cases with concurrent brain injury. The combined application of the three can provide a more comprehensive imaging basis for preoperative localization of epilepsy, helping to optimize surgical plans.

ELIGIBILITY:
Inclusion Criteria:

* with drug-resistant focal epilepsy defined by ILAE criteria
* Already performed 3.0 T epilepsy-protocol MRI and video-EEG
* Planned resective surgery or stereotactic EEG (SEEG) electrode implantation, and willingness to undergo all three PET scans: ¹⁸F-FDG, SV2A, and TSPO.
* Ability to understand study procedures and provide written informed consent.
* Availability of complete postoperative follow-up data with at least 12-month Engel outcome classification.

Exclusion Criteria:

-History of head trauma ,claustrophobia, rheumatic or autoimmune diseases, psychiatric disorders, severe somatic diseases (neurological,cardiovascular, etc.),previous heart or brain surgery, substance abuse, inability to refrain from hypnotics, magnetic implants, pregnancy, lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with drug-resistant focal epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value | 2 years
  Measures of specific binding of TSPO/SV2A/FDG
Standardized Uptake Value | 2 years
  Measures of specific binding of TSPO/SV2A/FDG measures of specific binding of the tracer